CLINICAL TRIAL: NCT02553525
Title: Effects of Stimulation Patterns of Deep Brain Stimulation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Emory University (Other); University of Florida (Other); Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00074235; R37NS040894 (NIH)
Record Dates: First submitted 2015-09-15; First posted 2015-09-17 (Estimated); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease; Essential Tremor; Multiple Sclerosis; Dystonia
Keywords: Deep Brain Stimulation; Movement Disorders; Parkinson Disease; Essential Tremor; Subthalamic Nucleus; Globus Pallidus; Thalamus; Tremor; Bradykinesia; Temporal Pattern; Electrical Stimulation; Neuromodulation; PD; ET; MS; STN; GPi; DBS; Nervous System Diseases; Neurodegenerative Diseases
MeSH Terms: conditions — Parkinson Disease; Essential Tremor; Multiple Sclerosis; Dystonia; Movement Disorders; Tremor; Hypokinesia; Nervous System Diseases; Neurodegenerative Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Stimulation Patterns (Experimental): This group will receive temporal patterns of stimulation that are designed to suppress oscillatory neural activity at theta- or beta-frequencies. These patterns are hypothesized to alleviate motor symptoms.
  Interventions: Procedure: Therapeutic Stimulation Patterns
- Symptogenic Stimulation Patterns (Experimental): This group will receive symptogenic patterns of stimulation that are designed to exacerbate oscillatory neural activity at theta- or beta-frequencies. These patterns are hypothesized to exacerbate motor symptoms.
  Interventions: Procedure: Symptogenic Stimulation Patterns

INTERVENTIONS:
Procedure: Therapeutic Stimulation Patterns — During deep brain stimulation (DBS) electrode implantation or implanted pulse generator (IPG) replacement surgery, different stimulation patterns that are designed to suppress oscillatory neural activity at theta- or beta-frequencies will be delivered in randomized order, and the subject will be blinded to the patterns. Neural activity and/or motor symptoms (tremor and/or bradykinesia) will be measured in response to DBS. Measurements will be made during 2- to 8-minute trials, in which stimulation will be off for the first half of the trial, and on for the remaining half. Neural activity and/or motor symptoms will be measured during both the off and on phases. The total amount of time necessary for data collection will be about 45 minutes.
  Arms: Therapeutic Stimulation Patterns
Procedure: Symptogenic Stimulation Patterns — During deep brain stimulation (DBS) electrode implantation or implanted pulse generator (IPG) replacement surgery, different stimulation patterns that are designed to exacerbate oscillatory neural activity at theta- or beta-frequencies will be delivered in randomized order, and the subject will be blinded to the patterns. Neural activity and/or motor symptoms (tremor and/or bradykinesia) will be measured in response to DBS. Measurements will be made during 2- to 8-minute trials, in which stimulation will be off for the first half of the trial, and on for the remaining half. Neural activity and/or motor symptoms will be measured during both the off and on phases. The total amount of time necessary for data collection will be about 45 minutes.
  Arms: Symptogenic Stimulation Patterns

SUMMARY:
The purpose of this study is to measure the effects of non-regular temporal patterns of deep brain stimulation (DBS) on motor symptoms and neural activity in persons with Parkinson's disease (PD), essential tremor (ET), dystonia or multiple sclerosis (MS). These data will guide the design of novel stimulation patterns that may lead to more effective and reliable treatment with DBS. These data will also enable evaluation of current hypotheses on the mechanisms of action of DBS. Improving our understanding of the mechanisms of action of DBS may lead to full development of DBS as a treatment for Parkinson's disease and may lead to future applications of DBS.

DETAILED DESCRIPTION:
This study will be conducted in the operating rooms at Duke University Medical Center, Emory University Hospital, University of Florida Shands Hospital or the UF Health Florida Surgical Center. The study will be performed during surgery on subjects who are undergoing implantation of the deep brain stimulation (DBS) system, or on subjects who are receiving surgical replacement of the implanted pulse generator (IPG) due to depleted batteries.

Subjects will receive temporary sterile extensions to the DBS electrode. These temporary extensions will connect to a stimulation and recording system and allow recording of neural activity. Over the course of ~45 minutes different non-regular temporal patterns of stimulation will be delivered unilaterally and the effects on neural activity and movement disorder symptoms will be measured. The stimulus waveform will be a charge-balanced biphasic pulse, with charge restricted to values below the limit set by the DBS IPG manufacturer, 30 μC/cm². After the study is completed, the temporary extensions will be removed, and the ordinary clinical conduct of the procedure will continue for treatment of the patient's movement disorder.

Tremor will be measured using an accelerometer in subjects with essential tremor (ET), multiple sclerosis (MS) and tremor-dominant Parkinson's disease (PD). Bradykinesia will be measured using a finger-tapping task on a computer mouse in subjects with Parkinson's disease who do not have dominant tremor symptoms. Subjects will be familiarized with the motor symptom evaluation tasks before surgery, and baseline measurements of tremor or bradykinesia may be recorded. Further, they may be asked to discontinue use of anti-parkinsonian and/or anti-tremor medications overnight prior to the study, to reduce variability of motor symptoms due to the time course of medications.

No general anesthesia will be given to subjects during surgery, and the procedure will be performed under local anesthesia to allow subjects to perform the tasks required in this study. Further, no sedation will be given to subjects receiving a replacement IPG, which can cause minor discomfort or anxiety in some patients. Subjects undergoing surgery for electrode implantation will receive monitored anesthesia care (MAC), in which sedation will be administered as needed, such that subjects are still responsive and pathological motor symptoms (tremor or bradykinesia) are present.

Following surgery, the subject's pre-operative MRI and post-operative high-resolution CT scans may be used to determine the location of DBS electrode contacts within the brain. However, participation in the study will not modify imaging procedures needed for standard care, and placement of the electrode during DBS implant surgery will not be altered by the research study.

There will be no additional costs to subjects as a result of being in this study. Additional operating room costs will be covered by institutional and/or grant resources.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's Disease (PD), Essential Tremor (ET) dystonia or Multiple Sclerosis (MS)
* Scheduled to undergo Deep Brain Stimulation (DBS) electrode implant, IPG implant or implanted pulse generator (IPG) replacement surgery
* Neurologically stable
* Able to understand the study and consent form

Exclusion Criteria:

* Inability to execute the motor tasks during the study
* Inability to tolerate withholding anti-parkinsonian and/or anti-tremor medications
* Clinically ineffective DBS

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-06-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Tremor Accelerometry | Day 1
  Tremor responses to deep brain stimulation (DBS) may be recorded by an accelerometer in subjects with essential tremor (ET), multiple sclerosis (MS) and tremor-dominant Parkinson's disease (PD). Tremor will be quantified by calculating the total power within a window of the power spectrum of the time series of the tremor, and this measure will be compared across stimulation patterns.
Bradykinesia Finger Tapping | Day 1
  Bradykinesia responses to deep brain stimulation (DBS) may be recorded by a computer mouse in subjects with Parkinson's disease (PD) who do not have dominant tremor symptoms. Bradykinesia will be quantified as the timing of alternating finger presses, a validated test of bradykinesia, and this measure will be compared across stimulation patterns.
Neural Activity | Day 1
  Neural activity consisting of electrically evoked compound action potentials (ECAPs), DBS local evoked potentials (DLEPs) and/or local field potentials (LFPs) may be recorded in response to deep brain stimulation (DBS). Neural activity characteristics will be compared across stimulation patterns and may be correlated with changes in severity of motor symptoms (tremor or bradykinesia).

SECONDARY OUTCOMES:
Electrode Location | Day 1
  Pre- and post-operative brain imaging obtained as part of standard care may be used to determine the location of subjects' implanted DBS electrode contacts. These data may be used to determine the location of the contacts used to record neural activity relative to the brain region targeted for stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Warren M Grill, PhD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - Emory University, Atlanta, Georgia
  - Duke University, Durham, North Carolina